CLINICAL TRIAL: NCT06401954
Title: Effects of High-Intensity Focused Electromagnetic Therapy Combined With Foot Core Training on Dynamic Foot Function in Individuals With Pronated Foot
Brief Title: High-Intensity Focused Electromagnetic Therapy Combined With Foot Core Training for Pronated Foot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202402010RINA
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Flexible Flatfoot
Keywords: pronated foot; foot core system; dynamic foot function; high-intensity focused electromagnetic therapy; foot core training
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIFEM with foot core training (Experimental): High-intensity focused electromagnetic therapy is used to stimulate intrinsic foot muscles, and foot core training is performed with intrinsic foot muscle isometric contraction exercise.
  Interventions: Device: High-intensity focused electromagnetic therapy; Behavioral: Foot core training
- HIFEM (Active Comparator): High-intensity focused electromagnetic therapy is used to stimulate intrinsic foot muscles
  Interventions: Behavioral: Foot core training
- Sham HIFEM with foot core training (Sham Comparator): Sham high-intensity focused electromagnetic therapy is applied on intrinsic foot muscles, and foot core training is performed with intrinsic foot muscle isometric contraction exercise.
  Interventions: Behavioral: Foot core training; Device: Sham high-intensity focused electromagnetic therapy

INTERVENTIONS:
Device: High-intensity focused electromagnetic therapy — High-intensity focused electromagnetic therapy is applied to intrinsic foot muscles, the intensity is set to stimulate muscle contraction.
  20 minutes of intervention, twice a week, and a total of 6 weeks
  Arms: HIFEM with foot core training
Behavioral: Foot core training — Foot core training will consist of 4 exercises with 10 repetitions per set and 3 sets per session for each exercise.
  Twice a week for a total of six weeks.
Device: Sham high-intensity focused electromagnetic therapy — Sham high-intensity focused electromagnetic therapy is applied to intrinsic foot muscles, the intensity is unable to stimulate muscle contraction.
  20 minutes of intervention, twice a week, and a total of 6 weeks
  Arms: Sham HIFEM with foot core training

SUMMARY:
The objective of this trial is to assess the effects of high-intensity focused electromagnetic therapy combined with foot core training targeting the intrinsic foot muscles on plantar load, static foot posture, intrinsic foot muscle morphology and intrinsic foot muscle activation in individuals with pronated foot.

The main questions it aims to answer are:

Question 1: To compare changes in plantar load following interventions of high-intensity focused electromagnetic therapy combined with foot core training, high-intensity focused electromagnetic therapy alone, and sham high-intensity focused electromagnetic therapy combined with foot core training.

Question 2: To compare changes in static foot posture, intrinsic foot muscle morphology, and intrinsic foot muscle activation following interventions of high-intensity focused electromagnetic therapy combined with foot core training, high-intensity focused electromagnetic therapy alone, and sham high-intensity focused electromagnetic therapy combined with foot core training.

Question 3: To assess the effects of each intervention on plantar load, static foot posture, intrinsic foot muscle morphology, and intrinsic foot muscle activation in individuals with pronated foot.

Participants will undergo stimulation of their intrinsic foot muscles through high-intensity focused electromagnetic therapy, and they will also be required to isometrically contract their intrinsic foot muscles during the designated exercise program. Researchers will assess the effects of high-intensity focused electromagnetic therapy combined with foot core training by evaluating plantar load during walking, static foot posture, intrinsic foot muscle morphology and intrinsic foot muscle activation during walking.

DETAILED DESCRIPTION:
The objective of this trial is to assess the effects of high-intensity focused electromagnetic therapy combined with foot core training targeting the intrinsic foot muscles on plantar load, static foot posture, intrinsic foot muscle morphology and intrinsic foot muscle activation in individuals with pronated foot.

The main questions it aims to answer are:

Question 1: To compare changes in plantar load following interventions of high-intensity focused electromagnetic therapy combined with foot core training, high-intensity focused electromagnetic therapy alone, and sham high-intensity focused electromagnetic therapy combined with foot core training.

Question 2: To compare changes in static foot posture, intrinsic foot muscle morphology, and intrinsic foot muscle activation following interventions of high-intensity focused electromagnetic therapy combined with foot core training, high-intensity focused electromagnetic therapy alone, and sham high-intensity focused electromagnetic therapy combined with foot core training.

Question 3: To assess the effects of each intervention on plantar load, static foot posture, intrinsic foot muscle morphology, and intrinsic foot muscle activation in individuals with pronated foot.

Eligible participants will be randomly assigned to one of three groups: the high-intensity focused electromagnetic therapy combined with foot core training group, the high-intensity focused electromagnetic therapy group, or the sham high-intensity focused electromagnetic therapy combined with foot core training group.

High-intensity focused electromagnetic therapy sessions will last for 20 minutes each, while the foot core training program will comprise 4 exercises, with 10 repetitions per set and 3 sets per session for each exercise. Participants will undergo these interventions twice a week over a 6-week period.

Plantar load and electromyographic signals of the abductor hallucis muscle during gait, ultrasonography for morphological analysis of the intrinsic foot muscles, and static foot posture will be evaluated at baseline and 6 weeks following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* Navicular drop test ≥ 10 mm
* Foot Posture Index ≥ 6
* Foot and ankle range of motion within normal limits

Exclusion Criteria:

* Rigid flatfoot
* Any congenital deformity of lower extremity
* Leg length discrepancy > 10 mm
* Lower extremity injuries or surgeries in recent 6 months
* Neurological deficits
* Contraindications of high-intensity focused electromagnetic therapy: pregnancy, unhealed wound, implanted electronic devices or other metal implants

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in plantar load at week 6 | baseline, week 6
  Plantar load is measured by in-shoe pressure measurement system, and the data is collected during walking.

SECONDARY OUTCOMES:
Change from baseline in static foot posture at week 6 | baseline, week 6
  Static foot posture is measured by navicular drop test and Foot Posture Index
Change from baseline in intrinsic foot muscle morphology at week 6 | baseline, week 6
  Intrinsic foot muscle morphology is measured by ultrasonography, include measurements of thickness of abductor hallucis, flexor hallucis brevis and flexor digitorum brevis, and cross-sectional area of abductor hallucis
Change from baseline in intrinsic foot muscle activation at week 6 | baseline, week 6
  Intrinsic foot muscle activation is measured by electromyography, and data is collected during walking

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, PhD, Principal Investigator — National Taiwan University, School of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Redmond AC, Crane YZ, Menz HB. Normative values for the Foot Posture Index. J Foot Ankle Res. 2008 Jul 31;1(1):6. doi: 10.1186/1757-1146-1-6. PMID 18822155
- [Background] Toullec E. Adult flatfoot. Orthop Traumatol Surg Res. 2015 Feb;101(1 Suppl):S11-7. doi: 10.1016/j.otsr.2014.07.030. Epub 2015 Jan 13. PMID 25595429
- [Background] Neal BS, Griffiths IB, Dowling GJ, Murley GS, Munteanu SE, Franettovich Smith MM, Collins NJ, Barton CJ. Foot posture as a risk factor for lower limb overuse injury: a systematic review and meta-analysis. J Foot Ankle Res. 2014 Dec 19;7(1):55. doi: 10.1186/s13047-014-0055-4. eCollection 2014. PMID 25558288
- [Background] Claus D, Waddy HM, Harding AE, Murray NM, Thomas PK. Hereditary motor and sensory neuropathies and hereditary spastic paraplegia: a magnetic stimulation study. Ann Neurol. 1990 Jul;28(1):43-9. doi: 10.1002/ana.410280109. PMID 2375632
- [Background] Razeghi M, Batt ME. Foot type classification: a critical review of current methods. Gait Posture. 2002 Jun;15(3):282-91. doi: 10.1016/s0966-6362(01)00151-5. PMID 11983503
- [Background] Buldt AK, Allan JJ, Landorf KB, Menz HB. The relationship between foot posture and plantar pressure during walking in adults: A systematic review. Gait Posture. 2018 May;62:56-67. doi: 10.1016/j.gaitpost.2018.02.026. Epub 2018 Feb 23. PMID 29524798
- [Background] Razak AH, Zayegh A, Begg RK, Wahab Y. Foot plantar pressure measurement system: a review. Sensors (Basel). 2012;12(7):9884-912. doi: 10.3390/s120709884. Epub 2012 Jul 23. PMID 23012576
- [Background] Cavanagh PR, Morag E, Boulton AJ, Young MJ, Deffner KT, Pammer SE. The relationship of static foot structure to dynamic foot function. J Biomech. 1997 Mar;30(3):243-50. doi: 10.1016/s0021-9290(96)00136-4. PMID 9119823
- [Background] Okamura K, Fukuda K, Oki S, Ono T, Tanaka S, Kanai S. Effects of plantar intrinsic foot muscle strengthening exercise on static and dynamic foot kinematics: A pilot randomized controlled single-blind trial in individuals with pes planus. Gait Posture. 2020 Jan;75:40-45. doi: 10.1016/j.gaitpost.2019.09.030. Epub 2019 Sep 29. PMID 31590069
- [Background] McKeon PO, Hertel J, Bramble D, Davis I. The foot core system: a new paradigm for understanding intrinsic foot muscle function. Br J Sports Med. 2015 Mar;49(5):290. doi: 10.1136/bjsports-2013-092690. Epub 2014 Mar 21. PMID 24659509
- [Background] Kelly LA, Cresswell AG, Racinais S, Whiteley R, Lichtwark G. Intrinsic foot muscles have the capacity to control deformation of the longitudinal arch. J R Soc Interface. 2014 Jan 29;11(93):20131188. doi: 10.1098/rsif.2013.1188. Print 2014 Apr 6. PMID 24478287
- [Background] Okamura K, Kanai S, Hasegawa M, Otsuka A, Oki S. The effect of additional activation of the plantar intrinsic foot muscles on foot dynamics during gait. Foot (Edinb). 2018 Mar;34:1-5. doi: 10.1016/j.foot.2017.08.002. Epub 2017 Aug 18. PMID 29175714
- [Background] Zhang X, Pauel R, Deschamps K, Jonkers I, Vanwanseele B. Differences in foot muscle morphology and foot kinematics between symptomatic and asymptomatic pronated feet. Scand J Med Sci Sports. 2019 Nov;29(11):1766-1773. doi: 10.1111/sms.13512. Epub 2019 Jul 26. PMID 31278774
- [Background] McKeon PO, Fourchet F. Freeing the foot: integrating the foot core system into rehabilitation for lower extremity injuries. Clin Sports Med. 2015 Apr;34(2):347-61. doi: 10.1016/j.csm.2014.12.002. Epub 2015 Jan 24. PMID 25818718
- [Background] Brijwasi T, Borkar P. A comprehensive exercise program improves foot alignment in people with flexible flat foot: a randomised trial. J Physiother. 2023 Jan;69(1):42-46. doi: 10.1016/j.jphys.2022.11.011. Epub 2022 Dec 14. PMID 36526555
- [Background] Huang C, Chen LY, Liao YH, Masodsai K, Lin YY. Effects of the Short-Foot Exercise on Foot Alignment and Muscle Hypertrophy in Flatfoot Individuals: A Meta-Analysis. Int J Environ Res Public Health. 2022 Sep 22;19(19):11994. doi: 10.3390/ijerph191911994. PMID 36231295
- [Background] Hara S, Kitano M, Kudo S. The effects of short foot exercises to treat flat foot deformity: A systematic review. J Back Musculoskelet Rehabil. 2023;36(1):21-33. doi: 10.3233/BMR-210374. PMID 35871320
- [Background] Utsahachant N, Sakulsriprasert P, Sinsurin K, Jensen MP, Sungkue S. Effects of short foot exercise combined with lower extremity training on dynamic foot function in individuals with flexible flatfoot: A randomized controlled trial. Gait Posture. 2023 Jul;104:109-115. doi: 10.1016/j.gaitpost.2023.06.013. Epub 2023 Jun 22. PMID 37379736
- [Background] Duncan D, Dinev I. Noninvasive Induction of Muscle Fiber Hypertrophy and Hyperplasia: Effects of High-Intensity Focused Electromagnetic Field Evaluated in an In-Vivo Porcine Model: A Pilot Study. Aesthet Surg J. 2020 Apr 14;40(5):568-574. doi: 10.1093/asj/sjz244. PMID 31665217
- [Background] Jacob C, Kinney B, Busso M, Chilukuri S, McCoy JD, Bailey C, Denkova R. High Intensity Focused Electro-Magnetic Technology (HIFEM) for Non-Invasive Buttock Lifting and Toning of Gluteal Muscles: A Multi-Center Efficacy and Safety Study. J Drugs Dermatol. 2018 Nov 1;17(11):1229-1232. PMID 30500146
- [Background] Silantyeva E, Zarkovic D, Astafeva E, Soldatskaia R, Orazov M, Belkovskaya M, Kurtser M; Academician of the Russian Academy of Sciences. A Comparative Study on the Effects of High-Intensity Focused Electromagnetic Technology and Electrostimulation for the Treatment of Pelvic Floor Muscles and Urinary Incontinence in Parous Women: Analysis of Posttreatment Data. Female Pelvic Med Reconstr Surg. 2021 Apr 1;27(4):269-273. doi: 10.1097/SPV.0000000000000807. PMID 31860567